CLINICAL TRIAL: NCT02745665
Title: A Pilot Case Control Study of Endothelial Function and Arterial Stiffness in Male Cyclists and Healthy Subjects
Brief Title: A Pilot Case Control Study of Vascular Function in Cyclists
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: St George's, University of London (Other)
Responsible Party: Sponsor
Other Study IDs: 16.0065
Record Dates: First submitted 2016-04-06; First posted 2016-04-20 (Estimated); Last update posted 2018-01-11 (Actual); Status verified 2018-01

CONDITIONS: Endothelial Function and Arterial Stiffness
MeSH Terms: interventions — Vascular Stiffness; Blood Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1-Elite Cyclist: 10 symptomatic cyclists with unilateral diagnosis of iliac EF,
  FLOW MEDIATED DILATION Ankle brachial pressure index (ABPI) PULSE WAVE VELOCITY AND AUGMENTATION INDEX Blood pressure RAMP Test
  Interventions: Other: flow mediated dilation (endothelial function); Other: ABPI; Other: Pulse wave velocity and augmentation index; Other: blood pressure; Other: ramp test
- 2-Amateur Cyclist: 10 asymptomatic cyclists with no evidence of EF
  FLOW MEDIATED DILATION ABPI PULSE WAVE VELOCITY AND AUGMENTATION Blood pressure RAMP Test
  Interventions: Other: flow mediated dilation (endothelial function); Other: ABPI; Other: Pulse wave velocity and augmentation index; Other: blood pressure; Other: ramp test
- 3-Control: 10 age-matched healthy male group
  FLOW MEDIATED DILATION ABPI PULSE WAVE VELOCITY AND AUGMENTATION Blood pressure RAMP Test
  Interventions: Other: flow mediated dilation (endothelial function); Other: ABPI; Other: Pulse wave velocity and augmentation index; Other: blood pressure; Other: ramp test

INTERVENTIONS:
Other: flow mediated dilation (endothelial function)
  Other Names: vascular function assessment
Other: ABPI
  Other Names: Duplex ultrasound and ankle brachial pressure index
Other: Pulse wave velocity and augmentation index
  Other Names: Arterial stiffness
Other: blood pressure
Other: ramp test
  Other Names: 20 minute static cycle ride to exhaustion

SUMMARY:
This is a pilot study with the purpose of measuring vascular function, assessed by evaluating arterial stiffness (pulse wave velocity and augmentation index) and endothelial function (flow mediated dilatation), in elite/amateur symptomatic male cyclists with unilateral Endofibrosis (EF), compared to asymptomatic males cyclists and to a group of age matched healthy males (non-athletes).

DETAILED DESCRIPTION:
Endofibrosis (EF) of the iliac arteries is a non-atheromatous flow-limiting condition specific to highly trained athletes. Although the pathophysiology is not well understood, haemodynamic injury and mechanical stress are considered to play a key role in developing EF. Recurrent exposure to these factors could trigger an arterial remodelling process that results in an intravascular lesion such as EF that more resembles an "adaptive intimal thickening". Although the natural history of this condition is not known, it is believed to be progressive with increasing numbers of reports of limb threatening ischaemia due to dissection and/or thrombosis of the arterial lumen. Therefore, it is imperative to understand the pathophysiological mechanism behind this condition in order to develop accurate diagnostic and screening criteria/tools for an early identification and characterization of EF. As there are no data in the literature supporting this hypothesis, the investigators have designed this pilot study to evaluate this hypothesis as to whether athletes with EF have evidence of vascular dysfunction in their arteries. There are currently no data on whether athletes who develop EF have underlying arterial disease or abnormalities. It is quite possible that people who develop EF have an underlying systemic endothelial dysfunction and that this may represent a risk factor for the development of the disease. Therefore the investigators will study non-invasively endothelial function (measured as flow mediated dilatation) as well as arterial stiffness (measured as pulse wave velocity and augmentation index) to improve the understanding about the structural and mechanical characteristics of the vascular tree in this cohort of patients.

ELIGIBILITY:
Inclusion Criteria:

* Males + 18 years elite or amateur racing cyclists with more than 3 years of training

Exclusion Criteria:

* - Subjects with a previous history of acute coronary syndrome (including myocardial infarction), stroke, transient ischaemic attack, cardiac surgery, other major cardiovascular (CV) surgery, or percutaneous coronary intervention (PCI), carotid surgery or carotid angioplasty, valvular heart, dysrhythmia
* subjects treated with cardiovascular medication for blood pressure, or cholesterol
* subjects with any clinical condition (diabetes, dyslipidaemia, obesity) that in the opinion of the investigator, may have a possible unfavourable effect on patient risk if included in the study, or is likely to interfere with the requirements of the study
* subject with characteristics that may interfere with adherence to the study protocol, such as dementia, substance abuse, history of non-compliance with prescribed medications, or medical appointment
* subject participating in another trial of an investigational drug or device within 30 days prior to screening will be excluded.
* subject that previously underwent surgery for iliac EF
* female subjects
* smokers

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Elite Cyclists with diagnosis of unilateral iliac EF - symptomatic Amateur racing cyclists with at least 3 years training asymptomatic Healthy males (age matched)
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-01-10 (Actual); Primary Completion 2018-06 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Flow Mediated Dilatation | 6 months
  is the gold standard to measure endothelial function with a High Definition Imaging 3000 ultrasound system (ATL, Bothell, WA, USA) equipped with a 12.5 MHz linear array transducer
pulse wave velocity | 6 months
  is the gold standard o assess arterial stiffness using the non invasive system of Complior (Arthec Medical)

SECONDARY OUTCOMES:
augmentation index | 6 months
  measurement to assess arterial stiffness using the non invasive system of Complior (Arthec Medical)

CONTACTS AND LOCATIONS:
Overall Officials: Rob Hinchliffe, Principal Investigator — St George's, University of London
Locations (1):
- St George's University Hospitals NHS Foundation Trust, Tooting, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Peach G, Schep G, Palfreeman R, Beard JD, Thompson MM, Hinchliffe RJ. Endofibrosis and kinking of the iliac arteries in athletes: a systematic review. Eur J Vasc Endovasc Surg. 2012 Feb;43(2):208-17. doi: 10.1016/j.ejvs.2011.11.019. Epub 2011 Dec 19. PMID 22186674